CLINICAL TRIAL: NCT05229029
Title: A Multicenter, Randomized, Double-blind Clinical Trial of TCM in Reducing CRF Caused by Chemotherapy in Cancer Patients
Brief Title: RSYR for Fatigue Reduction in Cancer Fatigue Caused by Chemotherapy
Acronym: TCM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Sun Hong, Director, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHEM FATI; SF2020-2-1023 (Other Grant/Funding Number: Beijing Science and Technology Commission)
Record Dates: First submitted 2021-12-03; First posted 2022-02-08 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Cancer-related Problem/Condition
Keywords: Chemotherapy; Fatigue; Cancer
MeSH Terms: conditions — Fatigue; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM decoction (Experimental): Compound granules of Traditional Chinese Medicine
  Interventions: Drug: TCM Formula
- placebo (Placebo Comparator): Placebo only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TCM Formula — TCM herbs：White peony 10g, angelica 10g, Astragalus 20g, Atractylodes macrocephala 10g, tangerine peel 6g, Poria cocos 10g, raw land 10g, cinnamon 3g, Polygala tenuifolia 6g, Schisandra chinensis 6g, raw licorice 6g.
  Other Names: RSYR decoction
  Arms: TCM decoction
Drug: Placebo — Mainly made of dextrin and caramel, containing 1/30 concentration of experimental group drugs
  Other Names: Placebo dicoction
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind clinical trial to evaluate the efficacy and safety of Chinese herbal compound in improving fatigue symptoms and quality of life in patients with chemotherapy.

DETAILED DESCRIPTION:
In this study, symptomatic indicators and quality of life were used as the main evaluation indicators. Patients with moderate to severe CRF who received dual drug chemotherapy were given traditional Chinese medicine compound and placebo intervention respectively. The data of fatigue symptoms, quality of life, sleep quality, blood routine test, liver and kidney function were observed and compared, so as to verify the traditional Chinese medicine compound prescription in improving the CRF symptoms and quality of life of chemotherapy patients validity.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor patients with pathological diagnosis
* Men and women aged 18-75
* KPS score ≥ 70, expected survival time more than 6 months
* The function of heart, lung, liver and kidney was normal
* Hemoglobin ≥ 8g
* Neuroendocrine function is normal
* BMI ≥ 18.5.
* Cancer pain, VAS score < 3
* Fatigue score ≥ 4
* syndrome differentiation is deficiency of Qi and blood

Exclusion Criteria:

* Brain metastases with Symptomatic
* Mental disease
* Severe infection
* Insomniacs
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue score | 21 days
  Self-assessed 24-hour fatigue symptom score. According to the NCCN fatigue guide, the score is 0-10 points, 0 points means no fatigue, 10 points means the most serious fatigue that can be imagined.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Sun, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No